CLINICAL TRIAL: NCT02307838
Title: Long-term Follow-up at 10 Years of Patients Enrolled in the Fingolimod Phase II Program in Relapsing Multiple Sclerosis (MS)
Brief Title: Long-term Follow-up of Fingolimod Phase II Study Patients
Acronym: ACROSS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CFTY720D2201E2
Record Dates: First submitted 2014-05-14; First posted 2014-12-04 (Estimated); Results first posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-02

CONDITIONS: Multiple Sclerosis, Relapsing Forms of Multiple Sclerosis
Keywords: Multiple Sclerosis, MS, RRMS, relapsing forms of multiple sclerosis, fingolimod, FTY720, Gilenya
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phase 2 CFTY720D2201 (NCT02307838) participants (Other): CFTY720D2201E2 participants did not receive any protocol specified treatment. The original D2201 study sites, who agreed to participate in this study, were required to locate their participants who were randomized in D2201 and asked them to return for a 10 year assessment, regardless of current treatment status.
  Interventions: Other: Assessments arm

INTERVENTIONS:
Other: Assessments arm — Protocol required assessments not provided in standard of care

SUMMARY:
This study collected follow-up data on approximately 90% of participants who were randomized and received one dose of study drug in FTY720D2201 (D2201). No study drug was given or required. Participants were required to be assessed at one or two visits, preferably at the original study site, but the option to be interviewed via phone or seen at home was provided. Information was gathered also on deceased participants. Assessments were performed only once within an 8 week period and included medical history, Multiple Sclerosis (MS) and Multiple Sclerosis Disease Modifying Therapy (MS DMT) history, Expanded Disability Status Scale (EDSS), Magnetic Resonance Imaging (MRI), and Multiple Sclerosis Functional Composite (MSFC).

DETAILED DESCRIPTION:
This was a multicenter follow-up study of patients originally enrolled in the Phase 2 D2201 study. Patients did not receive any protocol specified treatment. The original D2201 study sites who agreed to participate in this study were required to locate their patients who were randomized in Study D2201 and asked them to return for a 10-year assessment, regardless of their current treatment status. Locating the patient may have required the use of search and advertising strategies to find those patients currently lost to follow-up, in accordance with local privacy legislation. Patients currently being followed within Study FTY720D2399 (NCT01201356) were asked to participate in Study FTY720D2201E2 and if patients gave consent, were enrolled concurrently in both studies.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Randomized in study FTY720D2201 and received at least one dose of study drug.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (24):
- Canada (3):
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Denmark (2):
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Glostrup Municipality
- France (2):
  - Novartis Investigative Site, Marseille, France
  - Novartis Investigative Site, Lille
- Novartis Investigative Site, Würzburg, Germany
- Italy (4):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Gallarate, VA
- Novartis Investigative Site, Warsaw, Poland
- Portugal (2):
  - Novartis Investigative Site, Coimbra, Portugal
  - Novartis Investigative Site, Lisbon, Portugal
- Spain (6):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Valencia, Valencia
- Switzerland (2):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Zurich
- Novartis Investigative Site, Newcastle upon Tyne, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This extension study was a multicenter follow-up study of participants who enrolled in FTY720D2201 (NCT02307838). Although participants in this study did not receive study treatment, the participant flow is based on the treatments receive in FTY720D2201.
Pre-assignment Details: A total of 177 participants were enrolled into the study. However, 2 participants were erroneously enrolled into the study because they did not meet the inclusion criteria. Therefore, they were not included in any analyses, and as such, the participant flow is based on 175 participants.
Groups:
- FTY720 5.0 mg: In FTY720D2201, participants received FTY720 5.0 mg every day (q.d.) oral dose for 6 months.
- FTY720 1.25 mg: In FTY720D2201, participants received FTY720 1.25 mg q.d. oral dose for 6 months.
- Placebo: In FTY720D2201, participants received matching placebo to FTY720 q.d. for 6 months.
Period: Overall Study
Arm/Group | FTY720 5.0 mg | FTY720 1.25 mg | Placebo
Started | 56 | 64 | 55
Completed | 56 | 64 | 55
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: For baseline characteristics and analyses, participants were grouped according to FTY720 exposure: Continuous >= 8 years of FTY720 and Non-continuous < 8 years of FTY720. Non-continuous groups were broken down according to the high-efficacy DMTs' exposure. DMTs included natalizumab, mitoxantrone, alemtuzumab, rituximab, cladribine or ocrelizumab.
Groups:
- Continuous: Participants had exposure to FTY720 (study drug or commercially) for at least 8 years.
- Non-continuous: Participants had exposure to FTY720 (study drug or commercially) for less than 8 years.
- Non-continuous: Other DMTs: Participants had exposure to FTY720 (study drug or commercially) for less than 8 years. Also, participants were exposed to high-efficacy DMTs for less than 2 years. This group may have included participants who did not report any DMTs at all.
- Total: Total of all reporting groups
Arm/Group | Continuous | Non-continuous | Non-continuous: Other DMTs | Total
Number analyzed (Participants) | 104 | 16 | 55 | 175
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.4 (8.47) | 31.9 (9.05) | 38.9 (10.49) | 37.4 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 13 | 41 | 117
  Male | 41 | 3 | 14 | 58

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) in Expanded Disability Status Scale (EDSS)
Description: EDSS is a scale for assessing neurologic impairment in MS. It consists of eight functional systems (FS) which are used to derive the EDSS steps (score) ranging from 0 (normal) to 10 (death due to MS). The functional systems are Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel and Bladder, Cerebral and Other functions. Based on the assessment of each FS, the participant's score is determined between 0 to 10. A negative change from baseline indicates improvement.
Time Frame: baseline from core study (CFTY720D2201 (NCT00333138)), 10 years
Population: The full analysis set (FAS) included all participants who received at least one dose of study drug during FTY720D2201 and had at least one pre-treatment assessment in EDSS or magnetic resonance imaging (MRI) within study FTY720D2201.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Continuous | Non-continuous
Number analyzed (Participants) | 104 | 71
score on a scale | 0.58 (0.154) | 1.17 (0.185)
Statistical Analysis 1: Comparison: Continuous vs Non-continuous; Test type: Superiority or Other; p = 0.0155, ANCOVA; Difference in LS Means = -0.59, 95% CI 2-sided [-1.07 to -0.11]

2. Secondary Outcome: Number of Participants With Disability Progression
Description: Disability progression is defined as: 1.5-point increase from baseline in participants with baseline EDSS score = 0.0; OR 1-point increase in EDSS from baseline in participants with baseline EDSS score of 1.0 to 5.0 inclusive; OR 0.5-point increase in EDSS from baseline in participants with baseline EDSS score >5.0.
Time Frame: 10 Years
Population: The FAS included all participants who received at least one dose of study drug during FTY720D2201 and had at least one pre-treatment assessment in EDSS or magnetic resonance imaging (MRI) within study FTY720D2201.
Measure: Number; unit: Participants
Groups:
- Non-continuous: High Efficacy DMTs: Participants had exposure to FTY720 (study drug or commercially) for less than 8 years. Also, participants were exposed to high efficacy disease modifying therapies (DMTs) for at least 2 years.
Arm/Group | Continuous | Non-continuous: High Efficacy DMTs | Non-continuous: Other DMTs
Number analyzed (Participants) | 104 | 16 | 55
Participants | 35 | 8 | 29

3. Secondary Outcome: Number of Participants With EDSS <4 or <6
Description: EDSS is a scale for assessing neurologic impairment in MS. It consists of eight functional systems (FS) which are used to derive the EDSS steps (score) ranging from 0 (normal) to 10 (death due to MS). The functional systems are Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel and Bladder, Cerebral and Other functions. Based on the assessment of each FS, the participant's score is determined between 0 to 10. A positive change from baseline indicates improvement.
Time Frame: 10 years
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Continuous | Non-continuous: High Efficacy DMTs | Non-continuous: Other DMTs
Number analyzed (Participants) | 104 | 16 | 55
Participants
  EDSS <4 | 78 | 10 | 31
  EDSS <6 | 90 | 13 | 41

4. Secondary Outcome: Number of Participants Not Using a Wheelchair or Being Bedridden
Description: The number of participants not using a wheelchair or being bedridden was assessed.
Time Frame: 10 years
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Continuous | Non-continuous: High Efficacy DMTs | Non-continuous: Other DMTs
Number analyzed (Participants) | 104 | 16 | 55
Participants | 99 | 13 | 46

5. Secondary Outcome: Number of Participants Classified as Secondary Progressive MS (SPMS)
Description: SPMS follows an initial relapsing-remitting course. Most people who are diagnosed with relapsing-remitting multiple sclerosis (RRMS) will eventually transition to a secondary progressive course in which there is a progressive worsening of neurologic function (accumulation of disability) over time. Participants who were classified as SPMS were assessed.
Time Frame: 10 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Continuous | Non-continuous: High Efficacy DMTs | Non-continuous: Other DMTs
Number analyzed (Participants) | 104 | 16 | 55
Participants | 10 | 2 | 14

6. Secondary Outcome: Percentage of Participants With First Use of an Ambulatory Device
Description: First use of an ambulatory device was considered from EDSS 6.0 for participants having started FTY720D2201 (NCT00333138) with an EDSS score below 6.0.
Time Frame: 10 years
Population: The FAS was considered for the analysis. Only participants with evaluable data were included in the analysis. The FAS included all participants who received at least one dose of study drug during FTY720D2201 and had at least one pre-treatment assessment in EDSS or magnetic resonance imaging (MRI) within study FTY720D2201.
Measure: Number; unit: Percentage of participants
Arm/Group | Continuous | Non-continuous
Number analyzed (Participants) | 103 | 69
Percentage of participants | 12.4 | 17.6

7. Secondary Outcome: Percentage of Participants With First Use of a Wheelchair
Description: First use of a wheelchair was considered from EDSS 7.0 for participants having started FTY720D2201 (NCT00333138) with an EDSS score below 7.0.
Time Frame: 10 years
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Continuous | Non-continuous
Number analyzed (Participants) | 104 | 71
Percentage of participants | 4.9 | 16.9

8. Secondary Outcome: Change From Baseline in Multiple Sclerosis Fuctional Composite (MSFC) Component: Nine Hole Peg Test (9-HPT)
Description: The 9-HPT is a quantitative measure of upper extremity (arm and hand) function. Both the dominant and non-dominant hands are tested twice (two consecutive trials of the dominant hand, followed immediately by two consecutive trials of the non-dominant hand). The time limit per trial is 300 seconds. The right and left hand scores were the time in seconds it took to insert and remove 9 pegs ((the average scores from the four trials on the 9-HPT (the two trials for each hand are averaged, converted to the reciprocals of the mean times for each hand and then the two reciprocals are averaged)). A negative change from baseline indicates improvement.
Time Frame: baseline from core study, CFTY720D2201 (NCT00333138), 10 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Continuous | Non-continuous
Number analyzed (Participants) | 104 | 71
seconds | 2.29 (5.772) | 5.06 (14.523)

9. Secondary Outcome: Change From Baseline in MSFC Component: Paced Auditory Serial Addition Test (PASAT) Score
Description: The PASAT is a measure of cognitive function that specifically assesses auditory information processing speed and flexibility, as well as calculation ability. The PASAT is the last measure administered at each visit. It is presented on audio compact disc (CD) to control the rate of stimulus presentation. Single digits are presented every 3 seconds and the patient must add each new digit to the one immediately prior to it. The test result is the number of correct sums given (out of 60 possible). A positive change from baseline indicates improvement.
Time Frame: baseline from core study (CFTY720D2201 (NCT00333138)), 10 years
Population: The FAS was considered for the analysis. Only participants with both baseline and 10 year measurements were analyzed. The FAS included all participants who received at least one dose of study drug during FTY720D2201 and had at least one pre-treatment assessment in EDSS or magnetic resonance imaging (MRI) within study FTY720D2201.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Continuous | Non-continuous
Number analyzed (Participants) | 104 | 70
score on a scale | 0.54 (8.273) | -5.39 (12.428)

10. Secondary Outcome: Change From Baseline in MSFC Component: Timed 25-foot Walk Test Score
Description: The Timed 25-Foot Walk is a quantitative measure of lower extremity function. The patient is directed to one end of a clearly marked 25-foot (7.62 m) course and is instructed to walk 25 feet (7.62 meter) as quickly as possible, but safely. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task. The test scores were the time in seconds it took to walk the 25 feet. A negative change from baseline indicates improvement.
Time Frame: baseline from core study (CFTY720D2201 (NCT00333138)), 10 years
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Continuous | Non-continuous
Number analyzed (Participants) | 104 | 70
score on a scale | 1.32 (11.632) | 3.89 (16.070)

11. Secondary Outcome: Change From Baseline in Multiple Sclerosis Functional Composite (MSFC) Z Score
Description: MSFC is a composite measure encompassing information from the nine-hole peg test (arm dimension), timed 25 foot walk (leg dimension) and PASAT. The MSFC composite Z score was calculated as follows: (1) the average scores from the four trials on the 9-HPT (the two trials for each hand were averaged, converted to the reciprocals of the mean times for each hand and then the two reciprocals were averaged); (2) the average scores of two 25-Foot Timed Walk trials; (3) the number correct from the PASAT-3. The MSFC is based on the concept that scores for these three dimensions-arm, leg, and cognitive function are combined to create a single score (the MSFC) that can be used to detect change over time in a group of multiple sclerosis patients. This was done by creating Z-scores for each component of the MSFC, and averaging them to create an overall composite Z score.
Time Frame: baseline from core study (CFTY720D2201 (NCT00333138)), 10 years
Population: The FAS was considered for the analysis. Only participants with both baseline measurements for each MSFC component and 10 year measurements were analyzed. The FAS included all participants who received at least one dose of study drug during FTY720D2201 and had at least one pre-treatment assessment in EDSS or MRI within study FTY720D2201.
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Continuous | Non-continuous
Number analyzed (Participants) | 104 | 69
Z score | -0.11 (0.536) | -0.60 (1.297)

12. Secondary Outcome: Total Volume in T2 Lesion
Description: Total volume in T2 lesion was assessed by magnetic resonance imaging (MRI).
Time Frame: 10 years
Population: The FAS was considered for the analysis. Only participants with measurements at 10 years were included in the analysis. The FAS included all participants who received at least one dose of study drug during FTY720D2201 and had at least one pre-treatment assessment in EDSS or MRI within study FTY720D2201.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Continuous | Non-continuous
Number analyzed (Participants) | 98 | 54
mm^3 | 8685.4 (7743.05) | 11279.0 (12570.11)

13. Secondary Outcome: Change From Baseline in Total Volume of T2 Lesion
Description: Total volume in T2 lesion was assessed by magnetic resonance imaging (MRI). A negative change from baseline indicates improvement.
Time Frame: baseline from core study (CFTY720D2201 (NCT00333138)), 10 years
Population: The FAS was considered for the analysis. Only participants from the FAS who had both baseline and 10 years measurements were included in the analysis. The FAS included all participants who received at least one dose of study drug during FTY720D2201 and had at least one pre-treatment assessment in EDSS or MRI within study FTY720D2201.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Continuous | Non-continuous
Number analyzed (Participants) | 96 | 53
mm^3 | 1031.7 (3725.80) | 3636.7 (5259.84)

14. Secondary Outcome: Third Ventricle Diameter
Description: Third ventricle diameter was assessed by MRI.
Time Frame: 10 years
Population: The FAS was considered for the analysis. Only participants with 10 year measurements were analyzed. The FAS included all participants who received at least one dose of study drug during FTY720D2201 and had at least one pre-treatment assessment in EDSS or MRI within study FTY720D2201.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Continuous | Non-continuous
Number analyzed (Participants) | 97 | 56
mm | 5.28 (2.047) | 5.57 (2.648)

15. Secondary Outcome: Change From Baseline in Third Ventricle Diameter
Description: Third ventricle diameter was assessed by MRI. A negative change from baseline indicates improvement.
Time Frame: baseline from core study (CFTY720D2201 (NCT00333138)), 10 years
Population: The FAS was considered for analysis. Only participants who had both baseline and 10 year measurements were analyzed. The FAS included all participants who received at least one dose of study drug during FTY720D2201 and had at least one pre-treatment assessment in EDSS or MRI within study FTY720D2201.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Continuous | Non-continuous
Number analyzed (Participants) | 95 | 55
mm | 0.80 (0.848) | 0.92 (0.784)

16. Secondary Outcome: Percentage Brain Volume Change (PBVC)
Description: PVBC was assessed by MRI. A negative change from baseline indicates improvement.
Time Frame: baseline from core study (CFTY720D2201 (NCT00333138)), 10 years
Population: The FAS was considered for the analysis. Only participants with both baseline and 10 year measurements were analyzed. The FAS included all participants who received at least one dose of study drug during FTY720D2201 and had at least one pre-treatment assessment in EDSS or MRI within study FTY720D2201.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Continuous | Non-continuous
Number analyzed (Participants) | 85 | 48
Percent change | -9.28 (4.412) | -9.87 (2.909)

17. Secondary Outcome: Correlation Coeffcients Between FTY Treatment Duration and Disability Progression Parameters
Description: The correlation between FTY treatment duration and disability progression outcomes was assessed. The number presented in the table is the Pearson correlation coefficient, r.
Time Frame: 10 years
Population: The FAS was considered for the analysis. Only participants who had 10 year correlation measurements were analyzed. The FAS included all participants who received at least one dose of study drug during FTY720D2201 and had at least one pre-treatment assessment in EDSS or MRI within study FTY720D2201.
Measure: Number; unit: Pearson correlation coeffcient
Arm/Group | Continuous | Non-continuous
Number analyzed (Participants) | 104 | 71
Pearson correlation coeffcient
  EDSS score at year 10 (n=101,71) | -0.12 | -0.09
  Time to 1st use of a cane/crutch/walker (n=13,15) | 0.35 | 0.11
  Time to first documenting EDSS of >= 6.0 (n=12,11) | 0.27 | 0.00
  Time to first use of a wheelchair (n=5,12) | 0.57 | 0.33
  Time to first becoming bedridden (n=0,0) | NA — No participants had become bedridden. | NA — No participants had become bedridden.
  Time to first SPMS classification (n=10,16) | 0.38 | 0.32
  Year 10 PASAT-3 score (n=93,56) | -0.14 | 0.28
  Year 10 PASAT-3 score change from BL (n=93,56) | 0.01 | 0.39

ADVERSE EVENTS:
Groups:
- Non-continuous: High Efficacy DMTs: Participants had exposure to FTY720 (study drug or commercially) for less than 8 years. Also, participants were exposed to high-efficacy disease modifying therapies (DMTs) for at least 2 years.
Arm/Group | Continuous | Non-continuous: High Efficacy DMTs | Non-continuous: Other DMTs
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/16 | 0/55
Other Adverse Events (participants affected / at risk) | 0/104 | 0/16 | 1/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous (N=104) | Non-continuous: High Efficacy DMTs (N=16) | Non-continuous: Other DMTs (N=55)
Multiple sclerosis relapse (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.